CLINICAL TRIAL: NCT00898066
Title: Cytogenetic and Fluorescence In Situ Hybridization Studies in Multiple Myeloma
Brief Title: S0334 Analyzing Chromosomes in Patients With Newly Diagnosed Multiple Myeloma or Other Blood Disease
Status: Completed | Type: Observational
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: S0334; U10CA032102 (NIH); S0334 (Other: SWOG)
Record Dates: First submitted 2009-05-09; First posted 2009-05-12 (Estimated); Last update posted 2015-03-06 (Estimated); Status verified 2015-03

CONDITIONS: Lymphoma; Multiple Myeloma and Plasma Cell Neoplasm; Precancerous/Nonmalignant Condition
Keywords: Waldenstrom macroglobulinemia; monoclonal gammopathy of undetermined significance; primary systemic amyloidosis; stage I multiple myeloma; stage II multiple myeloma; stage III multiple myeloma
MeSH Terms: conditions — Lymphoma; Multiple Myeloma; Neoplasms, Plasma Cell; Precancerous Conditions; Waldenstrom Macroglobulinemia; Monoclonal Gammopathy of Undetermined Significance; Immunoglobulin Light-chain Amyloidosis | interventions — Cytogenetic Analysis; In Situ Hybridization, Fluorescence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Genetic: cytogenetic analysis — marrow and peripheral blood
Genetic: fluorescence in situ hybridization — marrow and peripheral blood

SUMMARY:
RATIONALE: Studying the chromosomes in samples of bone marrow and blood in the laboratory from patients with cancer or other blood diseases may help doctors learn more about the disease.

PURPOSE: This laboratory study is analyzing chromosomes in patients with newly diagnosed multiple myeloma or other blood disease.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the frequency of deletion 13 as detected by fluorescence in situ hybridization (FISH) and conventional cytogenetics in patients with newly diagnosed multiple myeloma (MM) or other monoclonal gammopathies (MG).
* Examine the prognostic value of specific subsets of chromosome aberrations detected by conventional cytogenetics and FISH in relation to event-free and overall survival in these patients.
* Compare the prognostic value of cytogenetics and FISH with other MM and MG prognostic factors in these patients.
* Correlate the presence of cytogenetic and FISH features with clinical pathophysiological, cellular, or other molecular characteristics in these patients.

OUTLINE: Patients receive treatment as directed by the treatment clinical trial on which they are registered. Patients undergo bone marrow or blood sample collection periodically for conventional cytogenetic analysis and fluorescence in situ hybridization studies (FISH). Samples are analyzed for deleted 13q/monosomy 13 and chromosomal abnormalities.

PROJECTED ACCRUAL: A total of 500 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of 1 of the following:

  * Multiple myeloma (MM)
  * Smoldering myeloma
  * Waldenstrom's macroglobulinemia (WM)
  * Monoclonal gammopathy of undetermined significance (MGUS)
  * Amyloidosis (AL)
* Newly diagnosed disease
* Must be currently registered, but have not begun therapy, on 1 of the following Southwest Oncology Group (SWOG) treatment clinical trials:

  * SWOG-S0115
  * SWOG-S0232
  * SWOG-S0340
  * All new SWOG coordinated MM, smoldering myeloma, WM, MGUS, or AL clinical trials activated on or after the activation date of this research study (SWOG-S0334)

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: pts from S0115, S0232, S0340, S0417 and all new SWOG MM SM, WM, MGUS studies after 9/1/05 before closure
Sampling Method: Non-Probability Sample
Enrollment: 37 (Actual)
Dates: Start 2005-09; Primary Completion 2007-06 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Frequency of deletion 13 as detected by fluorescence in situ hybridization (FISH) and conventional cytogenetics | 1 year
Prognostic value of specific subsets of chromosome aberrations detected by conventional cytogenetics and FISH in relation to event-free and overall survival | 1 year
Comparison of prognostic value of cytogenetics and FISH with other multiple myeloma and monoclonal gammopathy prognostic factors | 1 year
Correlation between the presence of cytogenetic and FISH features and clinical pathophysiological, cellular, or other molecular characteristics | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Diane L. Persons, MD, Study Chair — University of Kansas